CLINICAL TRIAL: NCT05177211
Title: A Phase 2 Study of Fedratinib in Myelodysplastic /Myeloproliferative Neoplasms (MDS/MPNs) and Chronic Neutrophilic Leukemia (CNL)
Brief Title: Fedratinib in Myelodysplastic /Myeloproliferative Neoplasms (MDS/MPNs) and Chronic Neutrophilic Leukemia (CNL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20963
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myeloproliferative Neoplasm; Chronic Neutrophilic Leukemia; MDS
Keywords: MPNs; CNL
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia, Neutrophilic, Chronic | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Fedratinib (Experimental): Participants will taken Fedratinib by mouth once a day every day of each 28 day cycle.
  Interventions: Drug: Fedratinib Pill

INTERVENTIONS:
Drug: Fedratinib Pill — Participants will be given Fedratinib at a dose of 400 mg PO once daily (4-100 mg capsules). Fedratinib can be given at any time during the day, but patients are advised to take the dose at the same approximate time every day.
  Other Names: Inrebic

SUMMARY:
The purpose of the study is to evaluate the effectiveness, safety, and tolerability of a study drug called fedratinib in participants with myelodysplastic/myeloproliferative neoplasms (MDS/MPNs) and chronic neutrophilic leukemia (CNL).

ELIGIBILITY:
Inclusion Criteria:

* Patient must understand and voluntarily sign an ICF prior to any study-related assessments/ procedures being conducted
* 18 years of age or older on day of signing informed consent.
* Morphologically confirmed diagnosis of one of the following in accordance with WHO (2016) diagnostic criteria:

  1. Atypical Chronic Myeloid Leukemia (aCML), BCR-ABL1 negative
  2. Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable (MDS/MPN-U)
  3. Myelodysplastic Syndrome/Myeloproliferative Neoplasm with ring sideroblasts and thrombocytosis (MDS/MPN-RS-T)
  4. Chronic Neutrophilic Leukemia (CNL).
* Palpable splenomegaly ≥ 5 cm below left costal margin (LCM), spleen volume ≥ 450 cc, AND/OR MPN-SAF TSS > 10.
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of 0, 1 or 2
* Able to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test at screening. A FCBP is considered when a sexually mature female: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months.
* A FCBP must agree to use of two methods of highly effective contraception, be surgically sterile, or abstain from heterosexual activity for the course of the study through 30 days after the last dose of study treatment.
* Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy. Men must agree to not donate sperm during study therapy and for 30 days after the last dose of study therapy

Exclusion Criteria:

* Any of the laboratory abnormalities as listed in the protocol.
* Patient is pregnant or lactating female
* Patient is a woman of childbearing potential as previously defined in inclusion #7, unless using effective contraception while on study treatment
* Patient is a man who is a partner with of a woman of childbearing potential, unless they agree to use effective contraception while on study treatment as previously defined in inclusion #9.
* Patient with prior history of encephalopathy, including Wernicke's Encephalopathy (WE)
* Patient has signs or symptoms of encephalopathy, including Wernicke's Encephalopathy (e.g., severe ataxia, ocular paralysis or cerebellar signs) in which case thiamine deficiency needs to be excluded and a brain MRI might be required to exclude possible Wernicke's encephalopathy
* Patient has thiamine deficiency if not corrected before enrollment on the study
* Patient with concomitant treatment with or use of pharmaceutical or herbal agents known to be moderate or strong inducers of CYP3A4 or dual CYP3A4 and CYP2C19 inhibitors. For a list of moderate or strong inhibitors or inducers of CYP3A4, see table 3-2 and 3-3 at https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers.
* Patient on any chemotherapy, immunomodulatory drug therapy (e.g., lenalidomide, pomalidomide, thalidomide, interferon-alpha), ruxolitinib, anagrelide, corticosteroids >10 mg/day prednisone or equivalent. Patients may remain on hydroxyurea (e.g., hydrea) if it is being employed to control leukocytosis as long as the patient has been on a stable dose for > 14 days prior to initiation of fedratinib.
* Prior treatment with fedratinib
* Patient on treatment with myeloid growth (e.g., G-CSF) factor within 14 days prior to initiation of fedratinib
* Patient on treatment with aspirin with doses > 150 mg daily.
* Patient with diagnosis of chronic liver disease (e.g., chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis).
* Patients with active (uncontrolled, metastatic) second malignancies are excluded.
* Patient with uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4).
* Patient with known human immunodeficiency virus (HIV), active infectious Hepatitis B (Hep B), and/or active Hepatitis C (Hep C).

  a. Patients with known HIV are eligible if the following criteria are met: i. Patient has CD4+ T-cell count ≥ 350 cells/µL ii. Patient is on established anti-retroviral therapy (ART) (with medications that are not specifically excluded due to potential interactions within this study) for at least four weeks prior to study enrollment and have an HIV viral load less than 400 copies/mL prior to enrollment.

  b. Patients with a history of Hep C infection are eligible if: i. Patient has completed curative antiviral treatment and has hepatitis C viral load below the limit of quantification ii. Pt has Hep C antibody positive but Hep C RNA negative due to prior treatment or natural resolution.
* Patient with serious active infection requiring IV anti-microbials.
* Patient with presence of any significant gastric or other disorder that would inhibit absorption of oral medication.
* Patient is unable to swallow capsules.
* Patient with participation in any study of an investigational agent (drug, biologic, device) within 30 days prior to start of fedratinib.
* Patient has any condition including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study.
* Patient has any condition that confounds the ability to interpret data from the study.
* Any major surgery or radiation therapy within four weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Objective Clinical Response Rate | Up to 24 weeks
  Response rate of fedratinib in MDS/MPN and CNL. Investigators will measure the proportion of patients achieving a clinical response from baseline to week 24 as defined by Complete Response (CR), Partial Response (PR) or Clinical Benefit (CB) by modified MDS/MPN IWG Proposed response criteria.

SECONDARY OUTCOMES:
Proportion of patients achieving spleen response at 12 weeks | at 12 weeks
  Participants spleen size will be measured and compared to baseline spleen size measurement. Spleen response is defined as 50% reduction in palpable splenomegaly of a spleen that is at least 10cm at baseline, a spleen that is palpable at more than 5 cm at baseline becoming non-palpable, or, in cases where volumetric evaluation is feasible, a ≥ 35% reduction in spleen volume in patients with a baseline spleen volume > 450 cc. Spleen responses by palpation will need to correlate with a 50% reduction in longest diameter of the spleen by imaging.
Proportion of patients achieving spleen response at 24 weeks | at 24 weeks
  Participants spleen size will be measured and compared to baseline spleen size measurement. Spleen response is defined as 50% reduction in palpable splenomegaly of a spleen that is at least 10cm at baseline, a spleen that is palpable at more than 5 cm at baseline becoming non-palpable, or, in cases where volumetric evaluation is feasible, a ≥ 35% reduction in spleen volume in patients with a baseline spleen volume > 450 cc. Spleen responses by palpation will need to correlate with a 50% reduction in longest diameter of the spleen by imaging.
Proportion of patients who have a 50% reduction in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score (MPN-SAF TSS) at 12 weeks | at 12 weeks
  Reduction in MPN-SAF TSS score will be measured by comparing TSS score at day 84 assessment to TSS score on cycle 1 day 1. Only patients with baseline TSS ≥ 10 will be eligible for symptom response. Patients who do not have a TSS score performed at day 84 assessment or who have discontinued study drug prior to day 84 assessment will be considered to not have 50% reduction in TSS.
  The MPN-SAF TSS is a questionnaire with nine items containing the most common symptoms reported by patients (concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss and fever), plus one item ("worst fatigue") from the "Brief Fatigue Inventory (BFI)". Each item has a score that ranges from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be). A higher score therefore indicates more severe symptoms
Proportion of patients who have a 50% reduction in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score (MPN-SAF TSS) at 24 weeks | at 24 weeks
  Reduction in MPN-SAF TSS score will be measured by comparing TSS score at day 84 assessment to TSS score on cycle 1 day 1. Only patients with baseline TSS ≥ 10 will be eligible for symptom response. Patients who do not have a TSS score performed at day 84 assessment or who have discontinued study drug prior to day 84 assessment will be considered to not have 50% reduction in TSS.
  The MPN-SAF TSS is a questionnaire with nine items containing the most common symptoms reported by patients (concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss and fever), plus one item ("worst fatigue") from the "Brief Fatigue Inventory (BFI)". Each item has a score that ranges from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be). A higher score therefore indicates more severe symptoms

OTHER OUTCOMES:
Patient's global impression of change (PGIC) at week 12 | at week 12
  Patient's global impression of change will be measured using the validated questionnaire wherein patients are asked about the change in their myelofibrosis symptoms since starting on the study. Patients can choose from one of seven potential answers: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. This will be reportedly qualitatively wherein the number of patients choosing particular answers will be tabulated and frequencies will be reported.
Patient's global impression of change (PGIC) at week 24 | at week 24
  Patient's global impression of change will be measured using the validated questionnaire wherein patients are asked about the change in their myelofibrosis symptoms since starting on the study. Patients can choose from one of seven potential answers: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. This will be reportedly qualitatively wherein the number of patients choosing particular answers will be tabulated and frequencies will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kuykendall, MD, Principal Investigator — Moffitt Cancer Center
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No